CLINICAL TRIAL: NCT06268899
Title: Evaluation of the Effectiveness of the Fırst Mobilization Protocol Developed for Knee Arthroplasty Patients
Brief Title: First Mobilization Protocol for Total Knee Arthroplasty Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Collaborators: Baskent University (Other)
Responsible Party: Principal Investigator, Sevil Güler, Professor, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: E-77082166-302.08.01-285977
Record Dates: First submitted 2024-02-09; First posted 2024-02-20 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Knee Arthroplasty
Keywords: Total Knee Arthroplasty; Nursing; Mobilization; Ambulation; First Mobilization Protocol; Orthopaedic and trauma nursing; Anxiety; Kinesiophobia; Mobilization related symptoms
MeSH Terms: conditions — Anxiety Disorders; Kinesiophobia

STUDY DESIGN:
Intervention Model Description: This study protocol describes the design of a single-center, single-blind, statistician-blind randomized controlled trial to be conducted in the Orthopedics and Traumatology Clinic of a provincial university hospital in Turkey.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant: the researcher learned the study and control groups after the pre-test data. The study group was trained with the mobilization protocol. The control group received training on the current mobilization procedure of the clinic. Participants did not know which group they were in.
  Outcomes Assessor. Study and control groups data were coded into the SPSS programme as group one and group two. Analysis of data was done by an independent statistician. The statistician has no information about which group the patients belong to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First mobilization protocol (Experimental): The protocol phases start one day before the patient's surgery and end on the first day of mobilization after surgery. The investigator explains the protocol steps to the patient before surgery and the patient is mobilized within the first 24 hours after surgery. Perform the protocol 4 times a day and more as tolerated. Mobilization protocol: Level 1: Patient is informed about mobilization and readiness is reinforced. Level 2: Passive and active ROM movements in bed should be performed at least 3 times a day. Level 3: Head of bed >60 degrees when the patient is sitting in bed. Duration target: 10-15 minutes. Level 4: Patient is seated on the edge of the bed. Duration target: 10-15 minutes. Level 5: The patient is helped to stand up. Level 6: First mobilization is achieved by allowing the patient to take 10-15 steps. The patient can mobilize at least 4 times a day.
  Interventions: Other: First mobilization protocol
- Control (No Intervention): No intervention was made to the control group, only data were collected at the same time as the study group.The patients in the control group was mobilized by the researchers according to the routine clinical mobilization practice.

INTERVENTIONS:
Other: First mobilization protocol — The protocol phases start one day before the patient's surgery and end on the first day of mobilization after surgery. The investigator explains the protocol steps to the patient before surgery and the patient is mobilized within the first 24 hours after surgery. Perform the protocol 4 times a day and more as tolerated. Mobilization protocol: Level 1: Patient is informed about mobilization and readiness is reinforced. Level 2: Passive and active ROM movements in bed should be performed at least 3 times a day. Level 3: Head of bed >60 degrees when the patient is sitting in bed. Duration target: 10-15 minutes. Level 4: Patient is seated on the edge of the bed. Duration target: 10-15 minutes. Level 5: The patient is helped to stand up. Level 6: First mobilization is achieved by allowing the patient to take 10-15 steps. The patient can mobilize at least 4 times a day.
  Arms: First mobilization protocol

SUMMARY:
This single blinded randomized controlled study evaluates the effect of developed First Mobilization Protocol applied to knee arthroplasty patients on state anxiety, kinesiophobia, initial mobilization related symptoms.

DETAILED DESCRIPTION:
Ensuring the mobilization of patients in the postoperative period, preventing complications resulting from inactivity, maintaining homeostatic balance and accelerating recovery are among the important goals of nursing care. For this reason, it is necessary to gradually increase the patients in line with the evidence-based data and the importance of mobilization should be emphasized. In this study, it was aimed to develop the first mobilization protocol for patients undergoing total knee arthroplasty and to evaluate the effectiveness of the developed protocol on patients' state anxiety, kinesiophobia, initial mobilization related symptoms.

The research is planned to be conducted in the Orthopedics and Traumatology Clinic of a university hospital in Turkey. The protocol of the study will be completed with78 patients who meet the sampling criteria (39 interventions, 39 controls), although it was designed as a single-center, single-blind randomized controlled and prospective study. Patient Information Form, State-Trait Anxiety Inventory, Tampa Kinesiophobia Scale and Initial Mobilization-Related Symptoms Evaluation Form will be used to collect the data of the study. Study; It is a single-center and single-blind randomized controlled experimental study protocol.

The data obtained within the scope of the study will be explained after being collected and analyzed. The effectiveness of the first mobilization protocol developed for tolal knee arthroplasty patients will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older,
* First time knee arthroplasty surgery,
* Have not received a diagnosis that will prevent communication,
* No physical disability,
* Mobilized during the implementation process of the research,
* Bilateral arthroplasty surgery is not performed,

Exclusion Criteria:

* Revision surgery performed,
* Patients who have undergone total hip or knee arthroplasty before,
* Inability to perform or delay mobilization due to complication(s) developed in the postoperative period,
* The patient cannot be mobilized on the first postoperative day (in the first 48 hours),
* Desire to leave the research voluntarily.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2023-01-08 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Anxiety evaluated using the Trait Anxiety Inventory (Trait Anxiety Inventory, TAI) | Change Trait Anxiety scale points on one day
  The "Trait Anxiety Inventory (STAI FORM TX-2, SDS)" allows the individual to express how he or she generally feels. the emotions and behaviors expressed in the scale items are according to their degrees; It is marked as (1) Almost Never, (2) Sometimes, (3) Often, and (4) Almost Always. 0-19 points from the scale mean no anxiety, 20-39 points mean mild, 40-59 points mean moderate, 60-79 points mean severe anxiety, and individuals with a score of 60 and above need professional help.
Kinesiophobia evaluated using the Tampa Kinesiophobia Scale | Change Kinesiophobia scale points on two days
  The Tampa Kinesiophobia Scale (TKS) was used to evaluate the patients' fear of moving. The scale consists of 17 items and has a Likert type feature. Scale items are used in the form of 4-point Likert scoring (1=Strongly disagree, 2=Disagree, 3=Agree, 4=Completely agree) and the total score ranges from 17-68. A high score from the scale indicates a high fear of movement. It is recommended to use the total score obtained from the scale in studies. It was stated that the test-retest reliability was 0.81.
Anxiety evaluated using the State Anxiety Inventory (State Anxiety Inventory, SAI) | Change Trait and State-Anxiety scale points on one day
  The State-Anxiety scale consists of twenty statements that evaluate how respondents' feel about anxiety "right now, at this moment" through four scales: one (not at all), two (somewhat), three (moderately so), and four (very much so). A rating of four indicates the presence of a high level anxiety and one indicates the absence of a high level anxiety. The anxiety level was found by calculation of scores, The range of scores is from 20-80, the higher the score indicating greater anxiety.
Symptoms evaluated using the Numerical Rating Scale for Symptoms Related to First Mobilization | Change symptoms points on one day
  Patients' symptoms related to the first mobilization (pain, dizziness, nausea, blackout, anxiety, stress, fear of damaging the surgery site, fear of falling, inability to walk/movement, walking distance on the first day, walking distance at the end of the first day, total walking at the end of the first day) distance, total mobilization per day, orthostatic intolerance, orthostatic hypotension) will be scored using a Numerical Comparison Scale from 0-10. This form will be used before and after mobilization on the day of the first mobilization of the patients.

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Gul ATAY DOYGACI, Master, Principal Investigator — Baskent Unversity
Locations (1):
- Gazi University Health Research and Application Center, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No